CLINICAL TRIAL: NCT04876456
Title: A Phase II Trial Evaluating the Efficacy of Cabozantinib in the Treatment of Incurable Patients With Refractory Germ Cell Tumors
Brief Title: A Phase II Trial of Cabozantinib With Patients With Refractory GCTs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer King (Other)
Collaborators: Exelixis (Industry); JDS Foundation Testis Cancer Clinical Trials Support Fund (Unknown)
Responsible Party: Sponsor-Investigator, Jennifer King, Assistant Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0752
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Germ Cell Tumor; Seminoma; Non-seminomatous Germ Cell Tumor; Ovarian Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Seminoma; Nonseminomatous germ cell tumor | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Patients will be treated with Cabozantinib 60mg orally daily continuously until disease progression, unacceptable toxicity, or trial closure.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Patients will be treated with Cabozantinib 60mg orally daily continuously until disease progression, unacceptable toxicity, or trial closure.

SUMMARY:
The purpose of the CTO-IUSCCC-0752 study is to investigate the use of Cabozantinib for patients with incurable, refractory germ cell tumors. Patients will be treated until evidence of disease progression, non-compliance with study protocol, unacceptable major toxicity, at subject's own request for withdrawal, or if the study closes for any reason.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Capable of understanding and complying with the protocol requirements.
3. Age ≥ 18 years at the time of consent.
4. Histological or serological evidence of germ cell tumor, including seminoma, non-seminoma, and women with ovarian GCTs.
5. Must have progressed after first-line cisplatin based combination chemotherapy AND demonstrated progression following at least one salvage regimen for advanced germ cell and now considered incurable with standard therapies, including further chemotherapy or surgery.

   5.1. "Failure" of prior therapy is defined as: 5.1.1. A >25% increase in the products of the perpendicular diameters of measurable tumor masses during prior therapy which are not amenable to surgical resection.

   5.1.2. The presence of new tumors that are not amenable to surgical resection 5.1.3. An increase in AFP or beta-hcg (two separate determinations at least one week apart are required if rising tumor markers are the only evidence of failure).

   NOTE: Subjects with clinically growing teratoma (normal declining tumor markers and radiographic or clinical progression) should be considered for surgery.
6. Subjects with relapsed primary mediastinal non-seminomatous germ cell tumor (PMNSGCT) are eligible
7. Subjects with late relapse (>2 years from previous chemotherapy) not amenable to resection are eligible if they have received first line platinum based chemotherapy and are deemed not amenable to surgical resection (no need for 1 salvage regimen in late relapse patients to be eligible).
8. Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
10. Adequate laboratory values obtained within 10 days prior to registration for protocol therapy and as defined below:

    10.1. Hemoglobin ≥9g/dL 10.2. WBC ≥2500/μL 10.3. Absolute neutrophil count ≥1500/mm3 10.4. Platelet count ≥100,000/mm3 10.5. Total bilirubin ≤1.5 X ULN except patients with documented Gilbert's syndrome (≤3 X ULN) 10.6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤3 X ULN; for patients with hepatic metastases, ALT and AST ≤5 X ULN; ALP ≤5 X ULN with documented bone metastases.

    10.7. Serum albumin ≥ 2.8 g/dl 10.8. (PT)/INR or partial thromboplastin time (PTT) test < 1.5x the laboratory ULN
    * This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or direct factor Xa inhibitors) should be on a stable dose.

    10.9. Serum creatinine ≤ 2.0 x ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation:

    a. Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72) b. Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85 10.10. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g
11. Female patients of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Prior treatment with Cabozantinib.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
3. Subjects who have not received ≥1 salvage treatment regimens (except late relapse) or have further potentially curative treatment options.
4. Known brain metastases or cranial epidural disease unless adequately treated and stable for at least 4 weeks prior to first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic at the time of first dose of study treatment.
5. Radiation therapy for bone metastasis within 2 weeks, or any other radiation therapy within 4 weeks prior to first dose of study treatment.
6. Expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
7. Treatment with investigational agent, any type of cytotoxic, biologic or other systematic anticancer therapy within 28 days prior to registration for protocol therapy.
8. Subjects with another active malignancy is not allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason < Grade 7 prostate cancers, or other cancer for which the subject has not required therapy for ≥1 year.
9. History of psychiatric illness or social situations that would limit compliance with study requirements.
10. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    10.1 Cardiovascular disorders:
    1. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    2. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    3. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.

10.c.1 Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation for at least 1 week before first dose of study treatment.

10.2 Gastrointestinal (GI) disorders associated with a high risk of perforation or fistula formation:

1. The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute Protocol Version Date: 03/08/2022 Page 17 obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
2. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

   Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.

   11. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.

   12. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.

   13. Lesions invading or encasing any major blood vessels. 14. Other clinically significant disorders that would preclude safe study participation per the investigator's opinion.

a. Serious non-healing wound/ulcer/bone fracture. b. Uncompensated/symptomatic hypothyroidism. c. Moderate to severe hepatic impairment (Child-Pugh B or C). 15. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.

16. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment.

Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

17. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.

   18. Pregnant or lactating females. 19. Inability to swallow tablets. 20. Previously identified allergy or hypersensitivity to components of the study treatment formulations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate | Start of the treatment until time of death or last follow up visit (up to 2 years)
  determined by the proportion of complete responses, partial responses, and stable disease for at least 3 months of therapy using RECIST 1.1 while including markers AFP/ beta-hcg.

SECONDARY OUTCOMES:
Objective response rate | Start of the treatment until time of death or last follow up visit (up to 2 years)
  Defined by proportion of complete response and partial response using RECIST 1.1 or tumor markers.
Overall survival | Start of the treatment until time of death or last follow up visit (up to 2 years)
  Measured by start of the treatment until time of death or last follow up visit.
Incidence of Adverse Events | Start of treatment until end of treatment safety assessments (up to 2 year)
  Toxicity measured by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and need for treatment delay, dose reduction, or early discontinuation.
Progression free survival | Start of the treatment until time of death or last follow up visit (up to 2 years)
  The start of the treatment until death or criteria for disease progression are met. Patients who are event-free (death or progression) at the time of data analysis will be censored at their last date of contact.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer King, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States